CLINICAL TRIAL: NCT00414375
Title: Early Versus Delayed Operation for Perforated Appendicitis With Abscess, a Pilot Study
Brief Title: Early Versus Delayed Operation for Perforated Appendicitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Shawn St. Peter, Children's Mercy Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06 11 164
Record Dates: First submitted 2006-12-19; First posted 2006-12-21 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 2009-03

CONDITIONS: Appendiceal Abscess
Keywords: Perforated Appendicitis; Abscess; Appendectomy
MeSH Terms: conditions — Appendicitis; Abscess | interventions — Drainage

ARMS (2):
- 1 (Active Comparator): Drainage with interval appendectomy
  Interventions: Procedure: Drainage and Interval Appendectomy
- 2 (Experimental): appendectomy on presentation
  Interventions: Procedure: Operation on Admission

INTERVENTIONS:
Procedure: Operation on Admission — Laparoscopic appendectomy on admission
  Arms: 2
Procedure: Drainage and Interval Appendectomy — drainage with interval appendectomy
  Arms: 1

SUMMARY:
The objective of this study is to scientifically evaluate two different operative strategies for perforated appendicitis with abscess.

The hypothesis is that the increased difficulty of early operation is balanced by the immense patient investment with delayed operation.

DETAILED DESCRIPTION:
This will be a single institution, prospective, randomized clinical trial involving patients who present to the hospital with perforated appendicitis with abscess. This will be a pilot study.

Power calculations are not used for a pilot study. One group will undergo a primary laparoscopic appendectomy. The other group will receive intravenous antibiotics with drainage if possible and a laparoscopic appendectomy 10 weeks after initiation of treatment at presentation. All 7 general pediatric surgeons will be involved with the operations, who are all comfortable with these management arms. The surgeon will not induce a significant confounding variable into this study. The laparoscopic appendectomy is approached in the same manner by all members of our group. Those named on the form are qualified by the IRB to obtain consent and/or will be accountable for overseeing the study.

Both groups will have the same antibiotic regiment. All data will be analyzed on intention-to-treat basis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with perforated appendicitis and an abdominal abscess diagnosed on CT scan.
* Children of any age will be included.

Exclusion Criteria:

* Patients with immune deficiency
* Another condition affecting surgical decision making or recovery (e.g. hemophilia, severe cardiac or respiratory co-morbidities).
* Acute sepsis or severe pain from perforation not allowing for delayed management.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2006-12; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Pilot | 3 months

SECONDARY OUTCOMES:
PIP and PedsQL4 scores, time to full feeds, days of hospitalization, recurrent abscess, number of recurrences, number of CT scans, operating time | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Shawn D St. Peter, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States